CLINICAL TRIAL: NCT05799768
Title: Ketogenic Diet Intervention in Patients With Rheumatoid Arthritis (RA): a Pilot Study
Brief Title: Ketogenic Diet in Rheumatoid Arthritis (RA)
Acronym: KETORA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Rheumatology Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020H0090
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis; Inflammation; Obesity; Ketogenic Dieting; Metabolic Syndrome
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation; Obesity; Metabolic Syndrome | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic diet plan (Experimental): Subjects will be provided extensive educational and ongoing support on the KD, including personalized coaching with the ability to text a dietitian at any time and expect a response within 12 hours. Diet adherence and progress will be assessed daily using at-home whole capillary blood ketone/glucose monitors, along with diet records. We will assess adherence based on days in ketosis following these parameters: (BHB ≥ 0.5mM). Adherence will be defined as > 80% of days in ketosis.
  Interventions: Behavioral: Ketogenic diet

INTERVENTIONS:
Behavioral: Ketogenic diet — Ketogenic diet counseling

SUMMARY:
This is a 6-week ketogenic diet (KD) intervention where participants with rheumatoid arthritis (RA) will follow a KD plan, supervised and monitored by a dietician. Participants will be provided extensive educational and ongoing support on the KD, including personalized coaching with the ability to text a dietitian at any time and expect a response within 12 hours. Diet adherence and progress will be assessed daily using at-home blood ketone/glucose monitors, along with diet records. Participants will fill out health related questionnaires and undergo assessments of body composition, RA disease activity. This study also includes blood draws and fat biopsy of the abdominal region.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA according to the ACR/EULAR 2010 criteria for RA.
* On stable doses of DMARDs and/ or biological agents (≥ 2 months prior to study enrollment)

Exclusion Criteria:

* Chronic inflammatory/ autoimmune disease other than RA (e.g. gout, inflammatory bowel disease such as Crohn's disease or ulcerative colitis, lupus, myositis, etc.)
* Prednisone or other glucocorticoid use in the last 4 weeks (exception: intra-articular glucocorticoid injections)
* Insulin use
* Hospitalization in the 30 days prior to study enrollment
* Acute or uncontrolled disease (e.g. cirrhosis, COPD, CKD)
* Malignancy
* Chronic infection (HIV, hep B/C, etc.)
* Heavy drinking
* On a ketogenic diet or exogenous ketone supplement (lses than 3 months prior to study enrollment)
* Recent weight loss (>5% in the last 2 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
hsCRP | 6 weeks
  Systemic marker of inflammation

SECONDARY OUTCOMES:
DAS28-CRP | 6 weeks
  RA disease activity measure

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided